CLINICAL TRIAL: NCT04177953
Title: Nivolumab With Chemotherapy in Pleural Mesothelioma After Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Bristol-Myers Squibb (Industry); Thoraxklinik Heidelberg gGmbH - Universitätsklinikum Heidelberg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICITA
Record Dates: First submitted 2019-11-11; First posted 2019-11-26 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pleural Mesothelioma Malignant
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; Pemetrexed; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carboplatin or Cisplatin and Pemetrexed (Active Comparator): Four cycles (q4w) platinum-based adjuvant chemotherapy i.v.:
  * carboplatin AUC5 or cisplatin 75 mg/m2
  * pemetrexed 500 mg/m2
  Interventions: Drug: Carboplatin AUC 5; Drug: Cisplatin 75 mg/m2; Drug: Pemetrexed 500 mg/m2
- Carboplatin or Cisplatin and Pemetrexed + Nivolumab (Experimental): Four cycles (q4w) of a combination of platinum-based adjuvant chemotherapy and immunotherapy i.v.:
  * carboplatin AUC5 or cisplatin 75 mg/m2
  * pemetrexed 500 mg/m2
  * nivolumab 480 mg flat-dose.
  Followed by up to 12 cycles (q4w) maintenance immunotherapy:
  - nivolumab 480 mg flat-dose i.v.
  Interventions: Drug: Carboplatin AUC 5; Drug: Cisplatin 75 mg/m2; Drug: Pemetrexed 500 mg/m2; Biological: Nivolumab Injection

INTERVENTIONS:
Drug: Carboplatin AUC 5 — chemotherapy iv
Drug: Cisplatin 75 mg/m2 — chemotherapy iv
Drug: Pemetrexed 500 mg/m2 — chemotherapy iv
Biological: Nivolumab Injection — Human monoclonal antibody
  Other Names: Opdivo
  Arms: Carboplatin or Cisplatin and Pemetrexed + Nivolumab

SUMMARY:
Patients with malignant pleural mesothelioma stage I-III who have undergone cytoreductive surgery with curative intend consisting of extended pleurectomy / decortication (eP/D) with or without hyperthermic intrathoracic chemoperfusion (HITOC) who will receive a maximum treatment duration of 16 cycles (4 cycles of chemotherapy in both arms + 12 cycles maintenance immunotherapy in treatment arm B). The main objective of the trial is Time-to-next-treatment (TNT), as well as safety and tolerability.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open-label study including patients with malignant pleural mesothelioma (MPM) in tumor stages I-III who have previously undergone cytoreductive surgery by extended pleurectomy/decortication with or without hyperthermic intrathoracic chemoperfusion (eP/D ± HITOC).

Patients who have histologically proven initial diagnosis of malignant pleural mesothelioma of epithelioid subtype (including biphasic histologic subtype identified during surgery), will be included in this study. Patients must have confirmed Eastern Cooperative Group (ECOG) status 0 to 2 as well to able to be included to the study.

Patients will be centrally randomized 1:1 to receive either platinum-based adjuvant chemotherapy iv (Arm A) or platinum-based adjuvant chemotherapy iv together with nivolumab (Arm B) and stratified to (HITOC (yes vs. no)), (ECOG (0,1 vs. 2)), (Result of prior resection (macroscopic complete vs incomplete resection) with macroscopic complete resection defined as residual amounts of tumor being less than 1 cm3.

Arm A (platinum-based adjuvant chemotherapy iv) patients randomized to Arm A will receive 4 cycles (q4w) chemotherapy i.v. (carboplatin AUC5 (area under curve) or cisplatin 75 mg/m2 and pemetrexed 500 mg/m2). Usually, pemetrexed is administered first as a 10 min infusion, followed by infusion of the platinum component (starting 30 min after pemetrexed infusion). Active treatment within this arm is limited to 4 months.

Arm B (platinum-based adjuvant chemotherapy iv) patients randomized to Arm B will receive 4 cycles (q4w) chemotherapy i.v. (carboplatin AUC5 (area under curve) or cisplatin 75 mg/m2 and pemetrexed 500 mg/m2) together with up to 12 cycles (q4w) maintenance immunotherapy with nivolumab iv (480mg fixed dose over 60 minutes). During cycles 1-4, when nivolumab is administered along with chemotherapy, nivolumab will be administered as the first infusion, followed by the chemotherapy components. Subjects may be dosed with nivolumab i.v. no less than 26 days from the previous dose of drug. Active treatment within this arm is limited to 16 cycles (4 cycles adjuvant combination therapy + 12 cycles maintenance immunotherapy).

Tumor tissue, blood and stool samples will be collected for accompanying research project. (Participation is optional for participant).

During treatment, clinical visits (blood cell counts, ECG, detection of toxicity) occur prior to every treatment dose. Safety of chemotherapy/nivolumab will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported.

During treatment, tumor response will be assessed by the Investigator according to modified RECIST for pleural lesions and RECIST 1.1 for non-pleural lesions (radiological imaging by CT and/or MRI of the chest and upper abdomen [including the entire liver and both adrenal glands] at 8 weeks (±7days) from the date of first drug administration, at 16 weeks (±7 days) and every 12 weeks (±7 days) thereafter, until the initiation of the next anti-cancer therapy or death. A post-End-of-Treatment anticancer therapy status (EOT and follow-up (FU)) as well as a Survival Status (follow-up (FU)) will be assessed 30 days-, 100 days- and every 12 weeks after End of Treatment (EOT).

ELIGIBILITY:
Inclusion Criteria:

1. Fully-informed written consent
2. Males and females ≥ 18 years of age
3. Histologically proven initial diagnosis of malignant pleural mesothelioma of epithelioid subtype (patients can also be included if biphasic histologic subtype has been identified during surgery)
4. Postoperative stage I-III (TNM 8th Edition; pT1-4, pN0-2, cM0). Patients are only included with a completeness of cytoreduction score (CC score) <3 (i.e., residual tumor thickness ≤2.5 cm).
5. Patients must have undergone cytoreductive surgery with curative intent consisting of extended pleurectomy/decortication (eP/D) ± hyperthermic intrathoracic chemotherapy (HITOC) performed
6. Surgery conducted ≤12 weeks (≤84 days) before study inclusion and patient recovered from post-surgical complications of eP/D or eP/D + HITOC
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
8. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial. Women must not be breastfeeding.
9. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
10. WOCBP must agree to follow instructions for method(s) of contraception for a period of 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo 5 half-lives. The terminal half-lives of nivolumab is approximately 25 days. WOCBP should use an adequate method to avoid pregnancy for approximately 5 months (30 days plus the time required for nivolumab to undergo 5 half-lives) after the last dose of investigational drug. Females must agree to refrain from egg donating (ova, oocytes) during the intervention period and for at least 5 months after last dose of study intervention.

Exclusion Criteria:

1. Metastatic disease.
2. Patients for which surgery was scheduled as a cytoreductive surgery with curative intent but was then defined as palliative P/D by the operating surgeon.
3. Previous drug therapy against MPM.
4. A continuous post-operative hospitalization > 6 weeks due to surgery-related complications.
5. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways.
6. Inadequate hematological, renal and hepatic functions including the following:

   1. WBC < 2,000/µL
   2. Neutrophils < 1,500/µL
   3. Platelets < 100 x 103/µL
   4. Hemoglobin <9.0 g/dL
   5. Serum creatinine >1.5 x ULN unless creatinine clearance ≥ 45 mL/min (measured or calculated using the Cockcroft-Gault formula). For application of cisplatin, creatinine clearance must be ≥ 60 mL/min. (measured or calculated using the Cockcroft-Gault formula).
   6. AST/ALT >3.0 x ULN
   7. Total bilirubin >1.5 x ULN (except subjects with Gilbert Syndrome who must have a total bilirubin level < 3.0 mg/dL)
7. Prior organ allograft or allogeneic bone marrow transplantation.
8. Concurrent or prior malignancy requiring or anticipated to require concurrent intervention.
9. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
10. Malignancies other than disease under study within 3 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).
11. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive study drug.
12. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or compliance with the study protocol.
13. Pregnant or breast-feeding women.
14. Positive testing for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
15. Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
16. Subjects with active, known, or suspected autoimmune disease. Subjects with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the medical monitor be consulted prior to signing informed consent.
17. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
18. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
19. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
20. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Time-to-next-treatment (TNT) assessed according to Kaplan-Meier analysis | From date of randomization, every 4 weeks up to 16 months until end of treatment
  Time-to-next-treatment (TNT) will be evaluated from time of randomization in order to assess efficacy of treatment, if addition of nivolumab to adjuvant chemotherapy and subsequent administration of nivolumab mono-agent as maintenance therapy will improve TNT.
Incidence and severity of adverse events according to CTC criteria | From date of randomization until 30 days after end of treatment
  Incidence and severity of adverse events according to CTC criteria

SECONDARY OUTCOMES:
Progression-free-survival (PFS): duration from the first study drug administration to the first documented evidence of disease progression or death of any cause | From date of randomization, every 4 weeks up to 16 months until end of treatment, and 30 days and 100 days post treatment and every 12 weeks during 32 weeks FU.
  Survival rates for the different time points will be determined using the Kaplan-Meier analysis and modified RECIST for MPM
Overall survival (OS) | From date of randomization, every 4 weeks up to 16 months until end of treatment, and 30 days and 100 days post treatment and every 12 weeks during 32 weeks FU.
  Survival rates will be assessed from randomization to death of any cause according to Kaplan-Meier analysis
Treatment Beyond Progression (TBP), duration of TBP in this population | From date of randomization until date of first documented progression or date of death from any cause, whichever came first, assessed during 16 months treatment, every 4 weeks, and 30 days and 100 days post treatment, every 12 weeks during 32 weeks FU.
  A descriptive analysis of the proportion of patients with Treatment Beyond Progression (TBP) as well as the duration of TBP within this population will be conducted. TBP is defined as the time of recording a tumor progression until initiation of any additional intervention against MPM due to disease progression (any systemic treatment; any locoregional measures [except for prophylactic radiotherapy to prevent procedure-track metastases]; any decision of the Investigator to switch the patient to BSC).
Patient reported outcomes: Quality of life (QoL, based on LCSS-Meso) | From date of Screening once and then after date of randomization every 4 weeks during treatment, up to 16 months and 30 days post treatment and every 12 weeks during 32 weeks FU.
  Questionnaires given to the patients (validated quality of life questionnaires LCSS-Meso (Lung Cancer Symptom Scale-Mesothelioma)).
  LCSS-Meso contains horizontal scales from best condition (maximum value/score = better outcome) to worst condition (minimum value/score = worse outcome), containing 8 questions regarding appetite, fatigue, cough, breathlessness, pain, lung disease complaints, lung disease complaint in terms of normal activities, and today´s quality of life.
Patient reported outcomes: Quality of life (QoL, based on EQ-5D) | From date of Screening once and then after date of randomization every 4 weeks during treatment, up to 16 months and 30 days post treatment and every 12 weeks during 32 weeks FU.
  Questionnaires given to the patients (validated quality of life questionnaires EQ-5D).
  EQ-5D contains questions in the field of mobility, self care, every day activities, pain, and prostration with fields to be ticked from best condition (maximum value/score = better outcome) to worst condition (minimum value/score = worse outcome). The questionnaire also contains a vertical scale of todays healthiness from 0 to 100 (0, 5, 15, 20... 95, 100). (0 = worst outcome, 100 = best outcome).
ECOG performance status | From date of Screening once and then after date of randomization every 4 weeks during treatment, up to 16 months until End of Treatment
  Eastern Cooperative Oncology Group patient performance status (Grading from 0 to 5)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Shah, MD, Principal Investigator — Thoraxklinik Heidelberg gGmbH, Medizinische Onkologie - Universitätsklinikum Heidelberg
Locations (12):
- Germany (12):
  - Vivantes Klinikum Neukölln, Klinik für Hämatologie, Onkologie und Palliativmedizin, Berlin
  - Klinikum Bremen Ost Pneumologie und Beatmungsmedizin, Bremen
  - Studienzentrum der Thorachirurgischen und Pneumologischen Klinik Klinken der Stadt Köln gGmbH Krankenhaus Merheim, Cologne
  - Ev. Kliniken Essen-Mitte, Klinik für Internistische Onkologie, Essen
  - Universitätsklinikum Freiburg Klinik für Innere Medizin I, Freiburg im Breisgau
  - Asklepios Fachklinik München-Gauting Thorakale Onkologie, Gauting
  - LungenClinic Grosshansdorf, Großhansdorf
  - Asklepios Klinikum Harburg, Klinik für Lungen-, Thorax und Atemwegserkrankungen, Harburg
  - Thoraxklinik Heidelberg gGmbH, Medizinische Onkologie, Heidelberg
  - Lungenklinik Hemer, Pneumologie und Thorakale Onkologie, Hemer
  - Universitätsklinikum Regensburg, Thoraxchirurgie, Regensburg
  - Robert-Bosch-Krankenhaus - Klinik Schillerhöhe, Onkologie, Stuttgart

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Shah R, Klotz LV, Chung I, Feisst M, Schneider MA, Riedel J, Bischoff H, Eichhorn ME, Thomas M. A Phase II Trial of Nivolumab With Chemotherapy Followed by Maintenance Nivolumab in Patients With Pleural Mesothelioma After Surgery: The NICITA Study Protocol. Clin Lung Cancer. 2021 Mar;22(2):142-146. doi: 10.1016/j.cllc.2020.10.005. Epub 2020 Oct 14. PMID 33158765